CLINICAL TRIAL: NCT00792142
Title: A Phase II Study of Maintenance Treatment With Sequential Bortezomib, Thalidomide and Dexamethasone Following Autologous Peripheral Blood Stem Cell Transplant in Patients With Multiple Myeloma
Brief Title: Bortezomib, Thalidomide, and Dexamethasone After Melphalan and Stem Cell Transplant in Treating Patients With Stage I-III Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06143; P30CA033572 (NIH); CHNMC-06143; MILLENNIUM-06143; CDR0000624513 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2008-11-14; First posted 2008-11-17 (Estimated); Results first posted 2020-09-17 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2020-01

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm; Neurotoxicity
Keywords: neurotoxicity; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell; Neurotoxicity Syndromes | interventions — Bortezomib; Dexamethasone; Melphalan; Thalidomide; Cytogenetic Analysis; In Situ Hybridization, Fluorescence; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (stem cell transplant, maintenance treatment) (Experimental): Patients receive high-dose melphalan IV over 30 minutes on days -2 and -1 and undergo autologous peripheral blood stem cell transplantation on day 0. Patients receive filgrastim IV or SC beginning on day 5 and continuing until blood counts recover. Beginning 4 to 8 weeks after transplantation, patients receive maintenance therapy comprising bortezomib IV on days 1, 8, and 15. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients also receive oral dexamethasone on days 1 to 4. Treatment with dexamethasone repeats every month for 12 months in the absence of disease progression or unacceptable toxicity. Beginning 2 weeks after completion of bortezomib, patients receive oral thalidomide once daily until disease progression.
  Interventions: Drug: bortezomib; Drug: dexamethasone; Drug: melphalan; Drug: thalidomide; Genetic: cytogenetic analysis; Genetic: fluorescence in situ hybridization; Other: laboratory biomarker analysis; Other: questionnaire administration; Procedure: autologous hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Drug: bortezomib — Given IV
Drug: dexamethasone — Given orally
Drug: melphalan — Given IV
Drug: thalidomide — Given orally
Genetic: cytogenetic analysis — Performed on baseline and post transplant bone marrow specimens
Genetic: fluorescence in situ hybridization — Performed on baseline and post transplant bone marrow specimens
Other: laboratory biomarker analysis — Baseline, post transplant and prior to start of bortezomib, every 3 months post transplant for the first year, after 6 cycles of bortezomib, every year after transplant for 2-4 years.
Other: questionnaire administration — Completed at baseline (within 6 weeks prior to enrollment) and at 2 months post transplant and once a month after that for the first year. For the second year the questionnaire will be completed every 3 months as long as on thalidomide for the duration of the study.
Procedure: autologous hematopoietic stem cell transplantation — Minimum dose of 2 X 10(6) CD34 + cells/kg day 0 after two days of treatment with Melphalan
Procedure: peripheral blood stem cell transplantation — Minimum dose of 2 X 10(6) CD34 + cells/kg day 0 after two days of treatment with Melphalan

SUMMARY:
RATIONALE: Bortezomib and thalidomide may stop the growth of multiple myeloma by blocking blood flow to the cancer. Bortezomib may also stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving bortezomib together with thalidomide and dexamethasone may kill any cancer cells that remain after high-dose melphalan and stem cell transplant in patients with multiple myeloma.

PURPOSE: This phase II trial is studying the side effects of giving bortezomib together with thalidomide and dexamethasone after melphalan and stem cell transplant and to see how well it works in treating patients with stage I-III multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the feasibility and toxicities of maintenance therapy with sequential bortezomib, thalidomide, and dexamethasone after high-dose melphalan and autologous peripheral blood stem cell transplantation in patients with multiple myeloma.
* To assess whether administration of sequential bortezomib, thalidomide, and dexamethasone can improve progression-free survival of these patients.

Secondary

* To assess whether administration of sequential bortezomib, thalidomide, and dexamethasone can increase complete remission rate and duration of response in these patients.
* To assess the impact of maintenance therapy with sequential bortezomib, thalidomide, and dexamethasone after transplantation on overall survival of these patients.
* To evaluate the influence of cytogenetic abnormalities (e.g., chromosome 13 deletion, 14 q32 abnormality, t [4;14], chromosome 1 q21 amplification, and chromosome 17 deletion) on outcome by performing conventional cytogenetic study and fluorescence in situ hybridization (FISH) studies on baseline and post-transplant bone marrow specimens.

OUTLINE:

* High-dose melphalan and autologous peripheral blood stem cell transplantation (PBSCT): Patients receive high-dose melphalan IV over 30 minutes on days -2 and -1 and undergo autologous PBSCT on day 0. Patients receive filgrastim (G-CSF) IV or subcutaneously beginning on day 5 and continuing until blood counts recover.
* Maintenance therapy: Beginning 4-8 weeks after transplantation, patients receive bortezomib IV on days 1, 8, and 15. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients also receive oral dexamethasone on days 1-4; treatment with dexamethasone repeats every month for 12 months in the absence of disease progression or unacceptable toxicity. Beginning 2 weeks after completion of bortezomib, patients receive oral thalidomide once daily until disease progression.

Patients complete the FACT-GOG neurotoxicity questionnaire periodically. Bone marrow samples are collected at baseline and post-transplant for cytogenetic analysis by FISH.

ELIGIBILITY:
Inclusion Criteria:

* Multiple Myeloma patients with symptomatic disease, stage II or III at diagnosis or progressive stage I requiring chemotherapy and/or radiation therapy (by Salmon-Durie classification), who are not eligible for tandem transplant study using TMI; because of previous radiation or eligibility criteria; documentation of disease staging by both Salmon-Durie classification and International Staging System (ISS) is required
* Patients with non-secretory myeloma should have measurable serum free-light chain protein by the Free-lite test or measurable disease such as a soft tissue myeloma
* A minimum of 4 x 10^6 of CD 34 Positive cell/kg has been harvested
* A Karnofsky performance status (KPS) of >= 70% is required unless the KPS is impaired due to bone disease
* No contraindication to the collection of a minimum of 4 x 10^6 CD34+ cells/kg by apheresis
* All patients must have signed a voluntary, informed consent in accordance with institutional and federal guidelines
* Bilirubin =< 1.5 mg/dl
* Serum glutamic oxaloacetic transaminase (SGOT) and serum glutamic pyruvate transaminase (SGPT) < 2.5 x upper limits of normal
* Creatinine clearance of >= 40cc/min
* Absolute neutrophil count of > 1000/ul
* Platelet count of > 100,000/ul
* Cardiac ejection fraction >= 45% by multigated acquisition (MUGA) scan and/or by echocardiogram
* Diffusing capacity of the lung for carbon monoxide (DLCO) >= 50% of predicted lower limit
* Human immunodeficiency virus (HIV) antibody tests negative
* No other medical, or psychosocial problems which in the opinion of the primary physician or principal investigator would place the patient at unacceptably high risk from this treatment regimen

Exclusion Criteria:

* Presence of peripheral neuropathy >= grade II
* Patients with evidence of disease progression (with >= 25% increase in M protein) on bortezomib and or thalidomide therapy prior to transplant
* Pregnant or nursing women, as well as women of child bearing age, who are unwilling to use a dual method of contraception and men who are unwilling to use condom
* Patients with history of hypersensitivity to bortezomib, boron or mannitol

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2008-01-16; Primary Completion 2014-04-21 (Actual); Study Completion 2014-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Firoozeh Sahebi, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Stem Cell Transplant, Maintenance Treatment): Patients receive high-dose melphalan IV 200mg/m^2 over 30 minutes on days -2 and -1 and undergo autologous peripheral blood stem cell transplantation (Minimum dose of 2 X 10(6) CD34 + cells/kg ) on day 0. Patients receive filgrastim 5ug/kg IV or SQ beginning on day 5 and continuing until blood counts recover. Beginning 4 to 8 weeks after transplantation, patients receive maintenance therapy comprising 1.3 mg/m^2 of bortezomib IV on days 1, 8, and 15. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients also receive 40mg of oral dexamethasone on days 1 to 4. Treatment with dexamethasone repeats every month for 12 months in the absence of disease progression or unacceptable toxicity. Beginning 2 weeks after completion of bortezomib, patients receive 50mg/day of oral thalidomide once daily until disease progression.
Period: Overall Study
Arm/Group | Treatment (Stem Cell Transplant, Maintenance Treatment)
Started | 45
Completed | 45
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Stem Cell Transplant, Maintenance Treatment)
Number analyzed (Participants) | 45
Age, Continuous [Median (Full Range); unit: years] | 55 [29 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 25
Region of Enrollment [Number; unit: participants]
  United States | 45

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: All grade 3 and above treatment-related adverse events (AEs) during bortezomib/dexamethasone treatment cycles.
Time Frame: After 4 months of maintenance therapy
Population: Five patients did not start the maintenance phase of the study because of neurotoxicity (n=3), thrombocytopenia (n=1), or withdrawal of consent (n=1).
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Stem Cell Transplant, Maintenance Treatment)
Number analyzed (Participants) | 40
Participants
  Leukopenia | 1
  Lymphopenia | 13
  Neutropenia | 2
  Thrombocytopenia | 1
  Cataract | 1
  Fatigue | 2
  Upper respiratory infection | 1
  Anxiety | 1
  Pain in extremity | 1
  Sinus bradycardia | 1
  Hyperglycemia | 4
  Hypophosphatemia | 3

2. Primary Outcome: One Year Overall Survival
Description: One year overall survival estimated using the product-limit method of Kaplan and Meier. Defined as the percentage of patients alive at year one after starting treatment.
Time Frame: From date of treatment initiation until death from any cause, assessed up to one year.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Stem Cell Transplant, Maintenance Treatment)
Number analyzed (Participants) | 45
percentage of participants | 95 [89 to 100]

3. Secondary Outcome: Count of Response in Patients Started on Maintenance Therapy
Description: Complete Response (CR): Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and < 5% plasma cells in bone marrow.
  Very Good Partial Response (VGPR): Serum and urine M-protein detectable by immunofixation but not on electrophoresis or 90% or greater reduction in serum M-protein plus urine M-protein level < 100mg per 24-h.
  Partial Response (PR): > 50% reduction of serum M-protein and reduction in 24-h urinary M-protein by > 90% or to < 200mg per 24-h In addition to the above listed criteria, if present at baseline, a . 50% reduction in the size of soft tissue plasmacytomas is also required.
  Stable Disease (SD): Not meeting criteria for CR, VGPR, PR or progressive disease.
  Relapse: Any of the following: Reappearance of serum or urine M-protein by immunofixation or electrophoresis Development of > 5% plasma cells in the bone marrow. Appearance of any other sign of progression (i.e., new plasmacytoma, lytic bone lesion)
Time Frame: Post-Thalidomide at 1 year.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Stem Cell Transplant, Maintenance Treatment)
Number analyzed (Participants) | 40
Participants
  CR | 20
  VPR | 2
  PR | 3
  Relapsed | 6
  Not Assessed | 9

4. Secondary Outcome: One Year Progression-free Survival (PFS)
Description: PFS estimated using the product-limit method of Kaplan and Meier. Defined as the percentage of patients progression-free at year one after starting treatment.
  International Myeloma Working Group uniform response criteria for disease progression:
  Increase of > 25% from baseline in Serum M-component and/or (the absolute increase must be > 0.5 g/dl); Urine M-component and/or (the absolute increase must be > 200 mg/24 h; Only in patients without measurable serum and urine M-protein levels:
  the difference between involved and uninvolved FLC levels. The absolute increase must be >l0mg/dl.
  Bone marrow plasma cell percentage: the absolute % must be > 10%C; Definite development of new bone lesions or soft tissue plasmacytomas.
  or definite increase in the size of existing bone lesions or soft tissue plasmacytomas Development of hypercalcemia (corrected serum calcium >11.5 mg/dl or 2.65 mmol/l) that can be attributed solely to the plasma cell proliferative disorder.
Time Frame: From start of treatment initiation until disease progression, relapse or death from any cause, assessed up to 1 year.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Stem Cell Transplant, Maintenance Treatment)
Number analyzed (Participants) | 45
percentage of participants | 88 [79 to 98]

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a period of 3 years and 11 months.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Treatment (Stem Cell Transplant, Maintenance Treatment)
Serious Adverse Events (participants affected / at risk) | 9/45
Other Adverse Events (participants affected / at risk) | 40/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Stem Cell Transplant, Maintenance Treatment) (N=45)
Myocardial ischemia (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Disease progression (General disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Peripheral nerve infection (Infections and infestations) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Vascular disorder (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Stem Cell Transplant, Maintenance Treatment) (N=45)
Hemoglobin decreased (Blood and lymphatic system disorders) | 31 (143)
Hemolysis (Blood and lymphatic system disorders) | 1 (1)
Lymphatic disorder (Blood and lymphatic system disorders) | 1 (2)
Palpitations (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 3 (4)
Ear disorder (Ear and labyrinth disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
External ear pain (Ear and labyrinth disorders) | 1 (1)
Hearing loss (Ear and labyrinth disorders) | 3 (10)
Tinnitus (Ear and labyrinth disorders) | 2 (2)
Cataract (Eye disorders) | 1 (3)
Dry eye syndrome (Eye disorders) | 1 (2)
Eye disorder (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 3 (3)
Watering eyes (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 5 (6)
Diarrhea (Gastrointestinal disorders) | 7 (8)
Dyspepsia (Gastrointestinal disorders) | 3 (6)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (2)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (2)
Lip pain (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (7)
Tooth disorder (Gastrointestinal disorders) | 1 (2)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (6)
Chest pain (General disorders) | 2 (3)
Chills (General disorders) | 1 (1)
Disease progression (General disorders) | 1 (1)
Edema limbs (General disorders) | 11 (12)
Fatigue (General disorders) | 15 (29)
Fever (General disorders) | 8 (9)
General symptom (General disorders) | 2 (2)
Injection site reaction (General disorders) | 1 (1)
Localized edema (General disorders) | 3 (3)
Pain (General disorders) | 3 (3)
Bladder infection (Infections and infestations) | 1 (1)
Bone infection (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Eye infection (Infections and infestations) | 2 (4)
Gastric infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 2 (2)
Mucosal infection (Infections and infestations) | 1 (1)
Opportunistic infection (Infections and infestations) | 1 (1)
Peripheral nerve infection (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 11 (16)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 15 (32)
Alkaline phosphatase increased (Investigations) | 8 (26)
Aspartate aminotransferase increased (Investigations) | 19 (38)
Bilirubin increased (Investigations) | 4 (4)
Carbon monoxide diffusing capacity decreased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 14 (41)
INR increased (Investigations) | 1 (1)
Leukocyte count decreased (Investigations) | 26 (103)
Lymphocyte count decreased (Investigations) | 22 (81)
Neutrophil count decreased (Investigations) | 22 (64)
Platelet count decreased (Investigations) | 20 (66)
Serum cholesterol increased (Investigations) | 6 (12)
Weight gain (Investigations) | 3 (8)
Weight loss (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 4 (5)
Blood glucose increased (Metabolism and nutrition disorders) | 17 (44)
Blood uric acid increased (Metabolism and nutrition disorders) | 4 (10)
Obesity (Metabolism and nutrition disorders) | 1 (2)
Serum albumin decreased (Metabolism and nutrition disorders) | 23 (57)
Serum calcium decreased (Metabolism and nutrition disorders) | 18 (36)
Serum calcium increased (Metabolism and nutrition disorders) | 6 (14)
Serum glucose decreased (Metabolism and nutrition disorders) | 15 (27)
Serum magnesium decreased (Metabolism and nutrition disorders) | 3 (4)
Serum magnesium increased (Metabolism and nutrition disorders) | 3 (6)
Serum phosphate decreased (Metabolism and nutrition disorders) | 9 (16)
Serum potassium decreased (Metabolism and nutrition disorders) | 12 (20)
Serum potassium increased (Metabolism and nutrition disorders) | 4 (5)
Serum sodium decreased (Metabolism and nutrition disorders) | 13 (28)
Serum sodium increased (Metabolism and nutrition disorders) | 2 (2)
Serum triglycerides increased (Metabolism and nutrition disorders) | 8 (16)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (20)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Buttock pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Joint disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 7 (16)
Kyphosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (5)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 3 (3)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 6 (12)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 (20)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 8 (11)
Facial muscle weakness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 10 (13)
Neuralgia (Nervous system disorders) | 1 (6)
Neurological disorder NOS (Nervous system disorders) | 1 (1)
Olfactory nerve disorder (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 33 (160)
Tremor (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 7 (10)
Depression (Psychiatric disorders) | 2 (4)
Insomnia (Psychiatric disorders) | 12 (24)
Hemoglobin urine positive (Renal and urinary disorders) | 2 (2)
Protein urine positive (Renal and urinary disorders) | 4 (5)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Vaginal dryness (Reproductive system and breast disorders) | 1 (1)
Vaginal inflammation (Reproductive system and breast disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (20)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccough (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (3)
Fat atrophy (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash desquamating (Skin and subcutaneous tissue disorders) | 13 (17)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 3 (5)
Flushing (Vascular disorders) | 3 (8)
Hematoma (Vascular disorders) | 1 (1)
Hemorrhage (Vascular disorders) | 1 (1)
Hot flashes (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 1 (2)
Hypotension (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-05-27): https://cdn.clinicaltrials.gov/large-docs/42/NCT00792142/Prot_SAP_000.pdf